CLINICAL TRIAL: NCT01557088
Title: Lp-PLA2, Progenitor Cells and Coronary Atherosclerosis in Humans
Brief Title: Lp-PLA2 and Coronary Atherosclerosis in Humans
Acronym: AIM 1 and II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Amir Lerman, Professor of Medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 08-008161; 5R01HL92954-01A1-05 (Other Grant/Funding Number: US NIH Grant); 1R01 AG31750-01A2-04 (Other Grant/Funding Number: NIA); 1R01AG031750-01A2 (NIH); 5R01HL092954 (NIH)
Record Dates: First submitted 2012-03-15; First posted 2012-03-19 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Coronary Atherosclerosis; Endothelial Dysfunction
Keywords: coronary artery disease; coronary artery spasm; small vessel coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease; Coronary Vasospasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Blood sampling from the Coronary Sinus and Aorta — Blood samples will be obtained from the aorta and the coronary sinus during the clinically scheduled angiogram and endothelial function testing.
Procedure: Intravascular Ultrasound of the coronary artery. — Intravascular Ultrasound will be completed for those subjects testing positive for coronary endothelial dysfunction during a clinically scheduled angiogram and endothelial function testing.

SUMMARY:
The majority of the acute coronary events are caused by coronary artery segments with minimal luminal disease, but with potentially significant vascular wall inflammation and oxidative stress leading to plaque vulnerability. It has become apparent that an initial injury at the endothelial surface, is the primary site of the mechanisms involved and a role for vascular inflammation and the interaction with oxidative stress continues to emerge. Lipoprotein-associated phospholipase A2 (Lp-PLA2) is a novel biomarker for vascular wall inflammation that circulates in the blood bound to both low density (LDL) and high density (HDL) lipoprotein and promotes vascular inflammation. Circulating levels of Lp-PLA2 mass and activity are an independent risk factor for cardiovascular events. Recent studies, demonstrating that Lp-PLA2 is also associated with coronary endothelial dysfunction. However, the relationship between Lp-PLA2 and early atherosclerotic changes in the coronary arteries, and the contribution of lipoprotein binding to the deleterious potential of Lp- PLA2 have not been elucidated. Our working hypothesis is that the endogenous local activation of the Lp-PLA2 pathway plays an integral role in early coronary atherosclerosis and contributes to the mechanism of coronary endothelial dysfunction and the structural and mechanical properties reflecting plaque vulnerability. Thus, the current application will characterize prospectively the correlation between the functional, mechanical, and structural vascular wall properties, and the systemic as well as the coronary activity of the Lp-PLA2 pathway.

DETAILED DESCRIPTION:
Aim I: Hypothesis: The extent of endothelial dysfunction will correlate with production of Lp-PLA2 and oxidative stress and correlates with the tissue characteristics of plaque vulnerability. The investigators will define the systemic and coronary gradient and production of markers of inflammation and oxidative stress and the presence of coronary endothelial dysfunction in patients with early coronary atherosclerosis.

Aim II: Hypothesis: The distribution of Lp-PLA2 on the LDL is associated with greater coronary endothelial dysfunction and correlates with the degree coronary atherosclerosis and plaque vulnerability. The investigators will define the distribution of Lp-PLA2 in patients with early coronary atherosclerosis and endothelial dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing coronary angiography including endothelial function testing
* male and female
* age 18 up to age 85

Exclusion Criteria:

* Heart failure with ejection fraction less that 40%
* unstable angina
* myocardial infarction or angioplasty within 6 months prior to entry into the study
* use of investigational agents within 1 month of entry into the study
* patients who require treatment with positive inotropic agents other than digoxin during the study
* patients with cerebrovascular accident within 6 months prior to entry into the study
* significant endocrine, hepatic or renal disorders
* local or systemic infectious disease within 4 weeks prior to entry into study
* pregnancy or lactation (women of child-bearing age will have a pregnancy test prior to angiogram)
* mental instability
* federal medical center inmates
* hemoglobin less than 12 mg/dL
* severe asthma

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2009-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Lp-PLA2 Assessment | baseline endothelial function assessment 6 months
  AIM 1: To assess the relationship between the 3 inflammatory measures of the Lp-PLA2 pathway (Lp-PLA2 mass, Lp-PLA2 activity and LysoPC) with endothelial function (as measured by the percent change in CAD (coronary artery disease) [Ach] and by the length of segments with endothelial dysfunction and plaque vulnerability (as measured by the necrotic core percent volume). AIM II: To assess the association between the percent of Lp-PLA2 residing on LDL and endothelial function (again measured by percent change in CAD [Ach], percent change in CBF (coronary blood flow)[Ach], and the length of endothelial dysfunction).

CONTACTS AND LOCATIONS:
Overall Officials: Amir Lerman, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States